CLINICAL TRIAL: NCT05226871
Title: A TREATMENT PROTOCOL FOR PARTICIPANTS CONTINUING FROM PFIZER-SPONSORED PALBOCICLIB CLINICAL STUDIES
Brief Title: Study for Participants Continuing From Pfizer-sponsored Palbociclib (a Study Medicine) Studies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5481173; 2021-005735-22 (EudraCT Number)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Head and Neck Cancer
Keywords: Hormone Receptor Positive Advanced Breast Cancer; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — palbociclib; Cetuximab; Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Other): Cetuximab
  Interventions: Drug: Cetuximab
- Arm 2 (Experimental): Palbociclib plus Cetuximab
  Interventions: Drug: Palbociclib; Drug: Cetuximab
- Arm 3 (Other): Palbociclib plus Fulvestrant
  Interventions: Drug: Palbociclib; Drug: Fulvestrant
- Arm 4 (Other): Palbociclib plus Letrozole
  Interventions: Drug: Palbociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — oral
  Other Names: IBRANCE
  Arms: Arm 2; Arm 3; Arm 4
Drug: Cetuximab — Intravenous (IV) infusion
  Arms: Arm 1; Arm 2
Drug: Fulvestrant — Intramuscular (IM)
  Arms: Arm 3
Drug: Letrozole — oral
  Arms: Arm 4

SUMMARY:
The purpose of this clinical trial is to provide study medicine(s) and learn about their safety. This study is seeking participants who:

* Have benefited from ongoing study treatment as determined by the study doctor in a Pfizer-sponsored palbociclib Parent Study
* Must agree to follow the reproductive criteria
* Are willing and able to comply with all scheduled visits, treatment plans, and other study procedures
* Can give signed informed consent documents

Participants in this study will continue to receive treatment as they were in the parent study. The time by which participants will take part in this study is retrospective (after completed parent study). We will examine the experiences of people receiving the study medicine(s). This will help us determine if the study medicine(s) are safe. During this time, the participants will be monitored for the safety of the study medicine(s).

DETAILED DESCRIPTION:
This is an open-label study to provide continued access to treatment for eligible participants who continue to derive clinical benefit as determined by the investigator from study intervention(s) in a Pfizer-sponsored palbociclib clinical study (Parent Study)

ELIGIBILITY:
Inclusion Criteria:

* Any participant who is receiving study treatment and deriving clinical benefit as determined by the investigator in a Pfizer-sponsored palbociclib Parent Study
* Participants must agree to follow the reproductive criteria
* Participants who are willing and able to comply with all scheduled visits, treatment plans, and other study procedures
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent document and protocol

Exclusion Criteria:

* Any medical reason that, in the opinion of the investigator or sponsor, precludes the participant from inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number/Percentage of Participants with Treatment-Emergent Adverse Events (AEs) Leading to Permanent Discontinuation of Study Treatment and Serious Adverse Events (SAEs) | Baseline up to 28 days after last dose of study intervention
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- UCSF Medical Center at Mission Bay, San Francisco, California, United States
- China (11):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
- Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
- Thailand (2):
  - Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok
  - Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkok
- Ukraine (3):
  - Regional Municipal Non-profit Enterprise "Bukovinian Clinical Oncology Center", Chernivtsi, Chernivetska Oblast
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipro
  - Municipal non-profit enterprise Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481173